CLINICAL TRIAL: NCT01682811
Title: Photodynamic Therapy for Benign Dermal Neurofibromas Using Levulan Kerastick For Topical Solution, Plus Illumination With Red Light
Brief Title: Phase I Photodynamic Therapy (PDT) for Benign Dermal Neurofibromas (NF1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Harry T Whelan, MD (Other)
Responsible Party: Sponsor-Investigator, Harry T Whelan, MD, Bleser Professor of Neurology, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO 14555
Record Dates: First submitted 2012-09-05; First posted 2012-09-11 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Neurofibromatoses
MeSH Terms: conditions — Neurofibromatoses | interventions — Percutaneous Collagen Induction; Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part 1 Levulan injection (Experimental): 5-aminolevulinic acid uptake by control lesions after Levulan vehicle (placebo) injection and 3 hr incubation, and by Levulan treated lesions after 3 or 24 hr incubation.
  Interventions: Drug: Part 1 Levulan injection
- Part 1 Levulan painting (Experimental): 5-aminolevulinic acid uptake by control lesions after Levulan vehicle (placebo) surface application and 3 hr incubation, and by Levulan treated lesions and 3 or 24 hr incubation.
  Interventions: Drug: Part 1 Levulan surface application
- Part 1 Levulan painted twice (Experimental): 5-aminolevulinic acid uptake by control lesions after Levulan vehicle (placebo) surface application twice or by Levulan treated lesions twice and 24 hr incubation.
  Interventions: Drug: Part 1 Levulan surface application twice
- Part 1 Levulan painted twice with microneedling (Experimental): 5-aminolevulinic acid uptake by control lesions after Levulan vehicle (placebo) surface application twice or by Levulan treated lesions twice and 24 hr incubation. All lesions prepared with microneedling.
  Interventions: Drug: Part 1 Levulan surface application twice with microneedling
- Part 2 Dose level 1 50 J/cm^2 (Experimental): Levulan (5-aminolevulinic acid) photodynamic therapy - Dose level 1 - 50 J/cm^2 633 nm red light to Levulan vehicle (placebo) treated control lesions or Levulan treated lesions and 24 hr incubation. Follow-ups on day 2 for punch biopsies, 14-28 days for evaluation of cutaneous adverse events, and every 3 months up to one year for lesion measurements.
  Interventions: Drug: Levulan (5-aminolevulinic acid) photodynamic therapy - Dose level 1
- Part 2 Dose level 2 100 J/cm^2 (Experimental): Levulan (5-aminolevulinic acid) photodynamic therapy - Dose level 2 - 100 J/cm^2 633 nm red light to Levulan vehicle (placebo) treated control lesions or Levulan treated lesions and 24 hr incubation. Follow-ups on day 2 for punch biopsies, 14-28 days for evaluation of cutaneous adverse events, and every 3 months up to one year for lesion measurements.
  Interventions: Drug: Levulan (5-aminolevulinic acid) photodynamic therapy - Dose level 2
- Part 2 Dose level 3 200 J/cm^2 (Experimental): Levulan (5-aminolevulinic acid) photodynamic therapy - Dose level 3 - 200 J/cm^2 633 nm red light to Levulan vehicle (placebo) treated control lesions or Levulan treated lesions and 24 hr incubation. Follow-ups on day 2 for punch biopsies, 14-28 days for evaluation of cutaneous adverse events, and every 3 months up to one year for lesion measurements.
  Interventions: Drug: Levulan (5-aminolevulinic acid) photodynamic therapy - Dose level 3

INTERVENTIONS:
Drug: Part 1 Levulan injection — Control or treatment lesions will be injected with Levulan vehicle only or active drug and incubated under occlusion for 3 or 24 hrs. A minimum of three lesions per group on the same subject will be treated. Lesions will then be excised in the normal manner, sectioned vertically, and checked for Protoporphyrin IX using fluorescence microscopy.
  Arms: Part 1 Levulan injection
Drug: Part 1 Levulan surface application — Control or treatment lesions will be painted with Levulan vehicle only or active drug, allowed to dry, and incubated under occlusion for 3 or 24 hrs. A minimum of three lesions per group on the same subject will be treated. Lesions will then be excised in the normal manner, sectioned vertically, and checked for Protoporphyrin IX using fluorescence microscopy.
  Arms: Part 1 Levulan painting
Drug: Part 1 Levulan surface application twice — Control or treatment lesions will be painted twice with Levulan vehicle only or active drug, allowed to dry between and after applications, and incubated under occlusion for 3 hrs. A minimum of three tumors per group on the same subject will be treated. Lesions will then be excised in the normal manner, sectioned vertically, and checked for Protoporphyrin IX using fluorescence microscopy.
  Arms: Part 1 Levulan painted twice
Drug: Part 1 Levulan surface application twice with microneedling — Control or treatment lesions will be prepared with microneedling, painted twice with Levulan vehicle only or active drug, allowed to dry between and after applications, and incubated under occlusion for 24 hrs. A minimum of three tumors per group on the same subject will be treated. Lesions will then be excised in the normal manner, sectioned vertically, and checked for Protoporphyrin IX using fluorescence microscopy.
  Arms: Part 1 Levulan painted twice with microneedling
Drug: Levulan (5-aminolevulinic acid) photodynamic therapy - Dose level 1 — 2-6 adult subjects with 3-8 lesions per (Levulan or control) group per subject. Controls will consist of lesions treated with vehicle only and light illumination, and will be paired with treatment lesions by the study doctor. Control lesions will be treated on the same subject as study lesions. Levulan will be incubated for 3-24 hours under occlusion, then gently rinsed with water and patted dry. Photoactivation of lesions treated with Levulan is then accomplished with 633 nm red light illumination. 633 nm light will be applied for 8 minutes to achieve a dose of 50 J/cm^2. There will be one treatment session per subject. Treatments will include a minimum of three test lesions and an additional three control lesions.
  Arms: Part 2 Dose level 1 50 J/cm^2
Drug: Levulan (5-aminolevulinic acid) photodynamic therapy - Dose level 2 — 2-6 adult subjects with 3-8 lesions per (Levulan or control) group per subject. Controls will consist of lesions treated with vehicle only and light illumination, and will be paired with treatment lesions by the study doctor. Control lesions will be treated on the same subject as study lesions. Levulan will be incubated for 3-24 hours under occlusion, then gently rinsed with water and patted dry. Photoactivation of lesions treated with Levulan is then accomplished with 633 nm red light illumination. 633 nm light will be applied for 16 minutes to achieve a dose of 100 J/cm^2. There will be one treatment session per subject. Treatments will include a minimum of three test lesions and an additional three control lesions.
  Arms: Part 2 Dose level 2 100 J/cm^2
Drug: Levulan (5-aminolevulinic acid) photodynamic therapy - Dose level 3 — 2-6 adult subjects with 3-8 lesions per (Levulan or control) group per subject. Controls will consist of lesions treated with vehicle only and light illumination, and will be paired with treatment lesions by the study doctor. Control lesions will be treated on the same subject as study lesions. Levulan will be incubated for 3-24 hours under occlusion, then gently rinsed with water and patted dry. Photoactivation of lesions treated with Levulan is then accomplished with 633 nm red light illumination. 633 nm light will be applied for 32 minutes to achieve a dose of 200 J/cm^2. There will be one treatment session per subject. Treatments will include a minimum of three test lesions and an additional three control lesions.
  Arms: Part 2 Dose level 3 200 J/cm^2

SUMMARY:
GENERAL OBJECTIVE The general objective is to assess the safety and efficacy of photodynamic therapy (PDT) in the treatment of neurofibromatosis 1 (NF1) tumors in the skin.

SPECIFIC OBJECTIVE This is a light dose escalation pilot study to determine the safety and efficacy of PDT using 5-aminolevulinic acid (ALA) and 633 nm light in the treatment of benign dermal neurofibromas.

Specifically, the primary goal of the current study is to determine the maximum tolerable light doses that can be administered to subjects undergoing topical photoillumination photodynamic therapy with standard application of Levulan Kerastick (ALA) for Topical Solution.

DETAILED DESCRIPTION:
STUDY DESIGN This protocol is a Phase I light dose escalation pilot study to determine the safety and, secondarily, the efficacy of PDT using Levulan and 633 nm light in the treatment of benign dermal neurofibromas. This protocol represents the first two parts of a planned three part study including both pediatric and adult subjects. Part 1 will consist of studying the penetration and uptake of the PS in neurofibromas that are scheduled for excision. These tumors will be excised for therapeutic reasons unrelated to this study, and so this study will place no further burden on the subject other than a 3-24 hr incubation of the Levulan on the tumor prior to excision. The primary hypothesis to be tested is whether Levulan will accumulate, and be converted to PpIX, by the tumor tissue more than by the surrounding normal tissue. Secondary hypotheses are that tumors incubated with Levulan will show greater fluorescence than untreated tumors and tumors incubated with vehicle only (placebo application).

As the Institutional Review Boards involved generally desire pilot data on adult populations first, we will with then proceed with the adult clinical trial portion of this protocol as part 2. Part 2 will use the optimum incubation time, if one has been identified in part 1, and add a dose escalation study of the amount of red light used to activate the Levulan. Part 3, with pediatric subjects, will commence at a future date, pending review of the initial adult study results.

ELIGIBILITY:
Inclusion Criteria:

Subjects with NF1 will be selected for photodynamic therapy on the following criteria.

1. Age: 18 years or older.
2. NF1 will be diagnosed by American Academy of Neurology guidelines.
3. Location of tumor: cutaneous, trunk or limbs only.
4. Tumor type: superficial dermal neurofibromas, less than or equal to 4 mm deep.
5. Growth confirmation: direct measurement for the dermal neurofibromas, ruler and photo-volumetric method.
6. Informed consent of subject.
7. Absence of any other malignancy.
8. Only failures to meet criteria 1-6 due to the primary disease will be disqualifying

Exclusion Criteria:

Subjects will be excluded from participation in the study on the basis of the following:

1. Life expectancy less than 1 year.
2. Pregnancy.
3. Inability to consent.
4. Cutaneous photosensitivity to the wavelengths used to activate PDT.
5. A diagnosis of porphyria.
6. Allergy to aminolevulinic acid or any of the Topical Solution Vehicle components.
7. Previous chemotherapy within 6 weeks of proposed PDT.
8. Other concurrent tumor therapy. -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03-12 (Actual); Primary Completion 2015-10-23 (Actual); Study Completion 2016-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry T Whelan, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- The Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Quirk B, Olasz E, Kumar S, Basel D, Whelan H. Photodynamic Therapy for Benign Cutaneous Neurofibromas Using Aminolevulinic Acid Topical Application and 633 nm Red Light Illumination. Photobiomodul Photomed Laser Surg. 2021 Jun;39(6):411-417. doi: 10.1089/photob.2020.4957. Epub 2021 Jan 20. PMID 33470897

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A prospective, controlled, nonrandomized phase I clinical trial was conducted between March 2012 and July 2016. This study included adult patients from Froedtert Hospital in Milwaukee, Wisconsin. NF1 patients were recruited through referral by their physician.
Units Other Than Participants: lesions
Groups:
- Experimental: Part 1 Levulan Painted Twice: 5-aminolevulinic acid uptake by control lesions after Levulan vehicle (placebo) surface application twice or by Levulan treated lesions twice and 24 hr incubation.
Period: Part 1 Levulan Injection
Arm/Group | Part 1 Levulan Injection | Part 1 Levulan Painting | Experimental: Part 1 Levulan Painted Twice | Part 1 Levulan Painted Twice With Microneedling | Part 2 Dose Level 1 50 J/cm^2 | Part 2 Dose Level 2 100 J/cm^2 | Part 2 Dose Level 3 200 J/cm^2
Started | 1; 9 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Control | 1; 3 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Treated 3 Hours | 1; 3 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Treated 24 Hours | 1; 3 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Completed | 1; 9 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Not Completed | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Period: Part 1 Levulan Painting
Arm/Group | Part 1 Levulan Injection | Part 1 Levulan Painting | Experimental: Part 1 Levulan Painted Twice | Part 1 Levulan Painted Twice With Microneedling | Part 2 Dose Level 1 50 J/cm^2 | Part 2 Dose Level 2 100 J/cm^2 | Part 2 Dose Level 3 200 J/cm^2
Started | 0; 0 lesions | 1; 9 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Control | 0; 0 lesions | 1; 3 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Treated 3 Hours | 0; 0 lesions | 1; 3 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Treated 24 Hours | 0; 0 lesions | 1; 3 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Completed | 0; 0 lesions | 1; 9 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Not Completed | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Period: Part 1 Levulan Painted Twice
Arm/Group | Part 1 Levulan Injection | Part 1 Levulan Painting | Experimental: Part 1 Levulan Painted Twice | Part 1 Levulan Painted Twice With Microneedling | Part 2 Dose Level 1 50 J/cm^2 | Part 2 Dose Level 2 100 J/cm^2 | Part 2 Dose Level 3 200 J/cm^2
Started | 0; 0 lesions | 0; 0 lesions | 2; 12 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Control | 0; 0 lesions | 0; 0 lesions | 2; 6 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Treated 24 Hours | 0; 0 lesions | 0; 0 lesions | 2; 6 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Completed | 0; 0 lesions | 0; 0 lesions | 2; 12 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Not Completed | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Period: Part 1 Levulan Paint Twice Microneedling
Arm/Group | Part 1 Levulan Injection | Part 1 Levulan Painting | Experimental: Part 1 Levulan Painted Twice | Part 1 Levulan Painted Twice With Microneedling | Part 2 Dose Level 1 50 J/cm^2 | Part 2 Dose Level 2 100 J/cm^2 | Part 2 Dose Level 3 200 J/cm^2
Started | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 2; 12 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Control | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 2; 6 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Treated 24 Hours | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 2; 6 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Completed | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 2; 12 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Not Completed | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Period: Part 2 Dose Level 1
Arm/Group | Part 1 Levulan Injection | Part 1 Levulan Painting | Experimental: Part 1 Levulan Painted Twice | Part 1 Levulan Painted Twice With Microneedling | Part 2 Dose Level 1 50 J/cm^2 | Part 2 Dose Level 2 100 J/cm^2 | Part 2 Dose Level 3 200 J/cm^2
Started | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 11; 60 lesions | 0; 0 lesions | 0; 0 lesions
Control | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 10; 30 lesions | 0; 0 lesions | 0; 0 lesions
Treated | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 10; 30 lesions | 0; 0 lesions | 0; 0 lesions
Completed | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Not Completed | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 11; 60 lesions | 0; 0 lesions | 0; 0 lesions
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 4 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 6 | 0 | 0
Period: Part 2 Dose Level 2
Arm/Group | Part 1 Levulan Injection | Part 1 Levulan Painting | Experimental: Part 1 Levulan Painted Twice | Part 1 Levulan Painted Twice With Microneedling | Part 2 Dose Level 1 50 J/cm^2 | Part 2 Dose Level 2 100 J/cm^2 | Part 2 Dose Level 3 200 J/cm^2
Started | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 3; 18 lesions | 0; 0 lesions
Control | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 3; 9 lesions | 0; 0 lesions
Treated | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 3; 9 lesions | 0; 0 lesions
Completed | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Not Completed | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 3; 18 lesions | 0; 0 lesions
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 3 | 0
Period: Part 2 Dose Level 3
Arm/Group | Part 1 Levulan Injection | Part 1 Levulan Painting | Experimental: Part 1 Levulan Painted Twice | Part 1 Levulan Painted Twice With Microneedling | Part 2 Dose Level 1 50 J/cm^2 | Part 2 Dose Level 2 100 J/cm^2 | Part 2 Dose Level 3 200 J/cm^2
Started | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Control | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Treated | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Completed | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Not Completed | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions

BASELINE CHARACTERISTICS:
Population: No subjects were enrolled into Part 2 Dose Level 3 as maximum tolerable dose had been established.
Units Other Than Participants: lesions
Groups:
- Experimental: Part 1 Levulan Injection: 5-aminolevulinic acid uptake by control lesions after Levulan vehicle (placebo) injection and 3 hr incubation, and by Levulan treated lesions after 3 or 24 hr incubation.
- Total: Total of all reporting groups
Arm/Group | Experimental: Part 1 Levulan Injection | Part 1 Levulan Painting | Part 1 Levulan Painted Twice | Part 1 Levulan Painted Twice With Microneedling | Part 2 Dose Level 1 50 J/cm^2 | Part 2 Dose Level 2 100 J/cm^2 | Part 2 Dose Level 3 200 J/cm^2 | Total
Number analyzed (Participants) | 1 | 1 | 2 | 2 | 11 | 3 | 0 | 20
Number analyzed (lesions) | 9 | 9 | 12 | 12 | 60 | 18 | 0 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 2 | 1 | 7 | 2 | 0 | 13
  >=65 years | 1 | 0 | 0 | 1 | 4 | 1 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2 | 8 | 1 | 0 | 13
  Male | 0 | 0 | 2 | 0 | 3 | 2 | 0 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    (all) |  |  |  |  |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2 | 2 | 11 | 3 |  | 20

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Photosensitizer Uptake and Conversion to Protoporphyrin IX
Description: The average fluorescence value for PpIX positive tumor areas in excised, sectioned tumors, as determined by fluorescence microscopy. PpIX signals were detected with excitation at 405 nm and emission with a 600 nm long pass filter. PpIX positive areas were determined to be those exhibiting fluorescence above background levels.
Time Frame: 24 hours
Population: The first participant contributed three lesions to each of the first three groups. The second participant likewise for the second three groups. The next two participants contributed three lesions each to each of the next two groups. The next two participants contributed likewise for the last two groups. PpIX positive areas were detected only in the last group.
Measure: Mean (Standard Deviation); unit: Densitometry units/micrometer squared
Units Other Than Participants: PpIX positive areas
Groups:
- Part 1 Levulan Injection Control Lesions: 5-aminolevulinic acid uptake by control lesions after Levulan vehicle (placebo) injection and 24 hr incubation.
- Part 1 Levulan Injection Treated Lesions 3 Hours: 5-aminolevulinic acid uptake by treated lesions after Levulan injection and 3 hr incubation.
- Part 1 Levulan Injection Treated Lesions 24 Hours: 5-aminolevulinic acid uptake by treated lesions after Levulan injection and 24 hr incubation.
- Part 1 Levulan Paint Control Lesions: 5-aminolevulinic acid uptake by control lesions after Levulan vehicle (placebo) surface application and 24 hr incubation.
- Part 1 Levulan Paint Treated Lesions 3 Hours: 5-aminolevulinic acid uptake by treated lesions after Levulan surface application and 3 hr incubation.
- Part 1 Levulan Paint Treated Lesions 24 Hours: 5-aminolevulinic acid uptake by treated lesions after Levulan surface application and 24 hr incubation.
- Part 1 Levulan Painted Twice Control Lesions: 5-aminolevulinic acid uptake by control lesions after Levulan vehicle (placebo) surface application twice and 3 hr incubation.
- Part 1 Levulan Painted Twice Treated Lesions: 5-aminolevulinic acid uptake by treated lesions after Levulan surface application twice and 3 hr incubation.
- Part 1 Levulan Painted Twice Control Lesions With Microneedling: 5-aminolevulinic acid uptake by control lesions after Levulan vehicle (placebo) surface application twice, on lesions prepared with microneedling, and 24 hr incubation.
- Part 1 Levulan Painted Twice Treated Lesions With Microneedling: 5-aminolevulinic acid uptake by treated lesions after Levulan surface application twice, on lesions prepared with microneedling, and 24 hr incubation.
Arm/Group | Part 1 Levulan Injection Control Lesions | Part 1 Levulan Injection Treated Lesions 3 Hours | Part 1 Levulan Injection Treated Lesions 24 Hours | Part 1 Levulan Paint Control Lesions | Part 1 Levulan Paint Treated Lesions 3 Hours | Part 1 Levulan Paint Treated Lesions 24 Hours | Part 1 Levulan Painted Twice Control Lesions | Part 1 Levulan Painted Twice Treated Lesions | Part 1 Levulan Painted Twice Control Lesions With Microneedling | Part 1 Levulan Painted Twice Treated Lesions With Microneedling
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 2 | 2
Number analyzed (PpIX positive areas) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
Densitometry units/micrometer squared |  |  |  |  |  |  |  |  |  | 304 (94)
Statistical Analysis 1: Comparison: Part 1 Levulan Painted Twice Treated Lesions With Microneedling; One-sample t-test comparing the absolute value to an alternate expected value of zero; Test type: Other; p = 0.0001, t-test, 1 sided

2. Primary Outcome: Part 2: Maximum Tolerated Dose (MTD) of 633 nm Red Light
Description: MTD was determined by testing increasing doses up to 200 J/cm^2 on dose escalation cohorts 1 to 3 with 3 to 6 participants each. MTD reflects the highest dose of red light that did not cause a Dose-Limiting Toxicity (DLT) in > 33% of participants. DLT was defined as pain during irradiation requiring cessation of the light treatment, or any serious cutaneous adverse events.
Time Frame: 48 hours
Population: Of the 14 enrolled in Part 2, 5 did not receive red light treatment per protocol. No subjects were enrolled in cohort 3 (200 J/cm^2) due to marked pain in cohort 2. In the opinion of the clinical dermatologist, higher dose levels would likely not be tolerable, and it would be unethical to escalate the light dose further. It was decided that the MTD would be set at 100 J/cm^2, and the highest dose level foregone.
Measure: Number; unit: joules/cm squared
Groups:
- All Participants: All participants who received at least 1 dose of 633 nm red light, either at 50 J/cm^2, 100 J/cm^2, or 200 J/cm^2.
Arm/Group | All Participants
Number analyzed (Participants) | 9
joules/cm squared | 100

3. Secondary Outcome: Part 1: Optimal Occlusion Time
Description: An optimal occlusion time may be apparent from the results of the three time points. If no optimal occlusion time is seen, any occlusion time from 3-24 hours may be chosen for part 2. This secondary outcome measure is not critical to continuing the study, but may be useful in guiding treatment protocols
Time Frame: 24 hours
Population: The first participant contributed three lesions to each of the first three groups. The second participant contributed three lesions to each of the second three groups. Only the six groups in the first two arms are relevant to this outcome measure.
Measure: Number; unit: hours
Units Other Than Participants: lesions
Arm/Group | Part 1 Levulan Injection Control Lesions | Part 1 Levulan Injection Treated Lesions 3 Hours | Part 1 Levulan Injection Treated Lesions 24 Hours | Part 1 Levulan Paint Control Lesions | Part 1 Levulan Paint Treated Lesions 3 Hours | Part 1 Levulan Paint Treated Lesions 24 Hours
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
Number analyzed (lesions) | 3 | 3 | 3 | 3 | 3 | 3
hours | NA — No optimal occlusion time was determined as no lesions showed PpIX fluorescence. | NA — No optimal occlusion time was determined as no lesions showed PpIX fluorescence. | NA — No optimal occlusion time was determined as no lesions showed PpIX fluorescence. | NA — No optimal occlusion time was determined as no lesions showed PpIX fluorescence. | NA — No optimal occlusion time was determined as no lesions showed PpIX fluorescence. | NA — No optimal occlusion time was determined as no lesions showed PpIX fluorescence.

4. Secondary Outcome: Part 2: Efficacy - Lesion Area Growth Rate
Description: Average lesion growth rates observed in ALA-treated lesions compared to vehicle-treated lesions within the same subjects.
Time Frame: 12 weeks
Population: Only 5 participants from Part 2 dose level 1 of the study had lesion sizes monitored during follow-up visits.
Measure: Mean (Standard Deviation); unit: millimeter squared/day post-treatment
Units Other Than Participants: lesions
Groups:
- Part 2 Dose Level 1 50 J/cm^2 Control: Levulan (5-aminolevulinic acid) photodynamic therapy - Dose level 1 - 50 J/cm^2 633 nm red light to Levulan vehicle (placebo) treated control lesions and 24 hr incubation. Follow-ups on day 2 for punch biopsies, 14-28 days for evaluation of cutaneous adverse events, and every 3 months up to one year for lesion measurements.
- Part 2 Dose Level 1 50 J/cm^2 Treated: Levulan (5-aminolevulinic acid) photodynamic therapy - Dose level 1 - 50 J/cm^2 633 nm red light to Levulan treated lesions and 24 hr incubation. Follow-ups on day 2 for punch biopsies, 14-28 days for evaluation of cutaneous adverse events, and every 3 months up to one year for lesion measurements.
Arm/Group | Part 2 Dose Level 1 50 J/cm^2 Control | Part 2 Dose Level 1 50 J/cm^2 Treated
Number analyzed (Participants) | 5 | 5
Number analyzed (lesions) | 14 | 14
millimeter squared/day post-treatment | 0.212 (0.364) | 0.081 (0.176)
Statistical Analysis 1: Comparison: Part 2 Dose Level 1 50 J/cm^2 Control vs Part 2 Dose Level 1 50 J/cm^2 Treated; Paired comparisons between treated and placebo lesions within subject; Test type: Other; p = 0.24, t-test, 2 sided

5. Secondary Outcome: Part 2: Cosmetic Improvement
Description: Potential cosmetic improvement using subject satisfaction scale.
Time Frame: 1 year
Population: No cosmetic improvement data was collected.
Groups:
- Part 2 Levulan (5-aminolevulinic Acid) Photodynamic Therapy.: Levulan (5-aminolevulinic acid) photodynamic therapy. 2-18 adult subjects with 3-8 lesions per (Levulan or control) group per subject. Controls will consist of lesions treated with vehicle only and light illumination, and will be paired with treatment lesions by the study doctor. Control lesions will be treated on the same subject as study lesions. Levulan will be incubated for 3-24 hours under occlusion, then gently rinsed with water and patted dry. Photoactivation of lesions treated with Levulan is then accomplished with 630 nm red light illumination. 630 nm light will be applied for varying periods of time in order to achieve a dose of 25, 50, or 100 J/cm2. There will be one treatment session per subject. Treatments will include a minimum of three test lesions and an additional three control lesions.
  Subjects will be seen at 24-48 hrs (48-72 hrs after Levulan application), and two weeks to one month after treatment at which times evaluation regarding dose toxicity will be made. Evaluations will include direct measurement of lesions, pain score, and cosmetic improvement (patient satisfaction).
  At the 2 day follow up visit, tumors will be punch biopsied, samples preserved in paraffin or formalin, and evaluated for cell death using TUNEL assays, H & E staining, or other methods.
Arm/Group | Part 2 Levulan (5-aminolevulinic Acid) Photodynamic Therapy.
Number analyzed (Participants) | 0

6. Secondary Outcome: Part 2: Pain Reduction
Description: Potential pain reduction, as measured by standard visual analog 1-10 scale.
Time Frame: 1 year
Population: No pain reduction data was collected.
Arm/Group | Part 2 Levulan (5-aminolevulinic Acid) Photodynamic Therapy.
Number analyzed (Participants) | 0

7. Post Hoc Outcome: TUNEL Assay.
Description: Average number of apoptotic cells per visual field among all TUNEL-evaluated lesion samples.
Time Frame: 48 hours
Population: Only 5 participants from Part 2 dose level 1 of the study had biopsies performed and lesions analyzed.
Measure: Mean (Standard Deviation); unit: apoptotic cells/visual field
Units Other Than Participants: Lesions
Arm/Group | Part 2 Dose Level 1 50 J/cm^2 Control | Part 2 Dose Level 1 50 J/cm^2 Treated
Number analyzed (Participants) | 5 | 5
Number analyzed (Lesions) | 15 | 5
apoptotic cells/visual field | 42.5 (19.9) | 1.1 (1.4)
Statistical Analysis 1: Comparison: Part 2 Dose Level 1 50 J/cm^2 Control vs Part 2 Dose Level 1 50 J/cm^2 Treated; Test type: Other; p = 0.002, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 weeks.
Groups:
- Part 1 Levulan (5-aminolevulinic Acid) Uptake.: Tumors will be incubated with Levulan or vehicle under occlusion for 3 or 24 hrs. A minimum of three tumors per treatment or control group will be treated on the same subject. Tumors will then be excised in the normal manner. Tumors will be sectioned vertically and checked for PpIX using fluorescence microscopy.
- Experimental: Part 2 Dose Level 1 50 J/cm^2: Levulan (5-aminolevulinic acid) photodynamic therapy - Dose level 1 - 50 J/cm^2 633 nm red light to Levulan vehicle (placebo) treated control lesions or Levulan treated lesions and 24 hr incubation. Follow-ups on day 2 for punch biopsies, 14-28 days for evaluation of cutaneous adverse events, and every 3 months up to one year for lesion measurements.
Arm/Group | Part 1 Levulan (5-aminolevulinic Acid) Uptake. | Experimental: Part 2 Dose Level 1 50 J/cm^2 | Part 2 Dose Level 2 100 J/cm^2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/11 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/11 | 0/3
Other Adverse Events (participants affected / at risk) | 0/6 | 1/11 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Levulan (5-aminolevulinic Acid) Uptake. (N=6) | Experimental: Part 2 Dose Level 1 50 J/cm^2 (N=11) | Part 2 Dose Level 2 100 J/cm^2 (N=3)
Skin burning with PDT - resolved (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — One participant in the first dose level cohort experienced pain upon red-light irradiation requiring cessation of PDT treatment. The pain resolved upon PDT cessation, with no sequelae.

LIMITATIONS AND CAVEATS:
No participants in part 2 completed 1 year of follow-up visits, and are reported as lost to follow-up. This necessarily limits all outcome measurements for part 2 other than the maximum tolerable dose measurement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No